CLINICAL TRIAL: NCT01189396
Title: A Randomized, Double- or Evaluator-blinded, Active- and Placebo-controlled, Cumulative-dose, Dose-escalating, Three-arm, Cross-over Study, in 24 Asthma Patients
Brief Title: Escalating and Cumulative-Dose Study of Pharmacokinetics (PK), Pharmacodynamics (PD) and Safety of A006
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amphastar Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: API-A006-CL-C
Record Dates: First submitted 2010-08-24; First posted 2010-08-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Asthma; Bronchospasm; Chronic Obstructive Pulmonary Disease (COPD)
Keywords: asthma; bronchospasm; COPD; reversibility; efficacy
MeSH Terms: conditions — Asthma; Bronchial Spasm; Pulmonary Disease, Chronic Obstructive | interventions — OIC-A006; Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- T (Experimental): Four doses of A006 taken in 30 minute intervals. Doses will have an escalating number of inhalations (1, 1, 2, and 4 inhalations). Total cumulative Albuterol dose at 90 minutes is 1440 mcg.
  Interventions: Drug: A006
- R (Active Comparator): Four doses of Proventil-HFA taken in 30 minute intervals. Doses will have an escalating number of inhalations (2, 2, 4, and 8 inhalations). Total cumulative Albuterol dose at 90 minutes is 1440 mcg.
  Interventions: Drug: Proventil-HFA
- P (Placebo Comparator): Four doses of Placebo DPI taken in 30 minute intervals. Doses will have an escalating number of inhalations (1, 1, 2, and 4 inhalations). Total cumulative Albuterol dose at 90 minutes is 0 mcg.
  Interventions: Drug: Placebo DPI

INTERVENTIONS:
Drug: A006 — Albuterol DPI with 180 mcg Albuterol/inhalation
  Arms: T
Drug: Placebo DPI — Placebo DPI with 0 mcg Albuterol/inhalation
  Arms: P
Drug: Proventil-HFA — Albuterol MDI with 90 mcg Albuterol/inhalation
  Arms: R

SUMMARY:
The main objective is to evaluate the bronchodilatory efficacy, safety and pharmacokinetic profiles of A006 (Albuterol Dry Powder Inhaler (DPI)), in comparison with those of an active control, Proventil-HFA (Albuterol Metered Dose Inhaler (MDI)), and a Placebo DPI in escalating and cumulative-doses up to 1440 mcg, eight (8) times of the proposed clinical dose.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥ 50 kg for men and ≥ 45 kg for women, and BMI within the range of 18.5 - 30.0 kg/m2 inclusive;
* Sitting blood pressure ≤ 135/90 mmHg;
* Demonstrating negative alcohol/drug screen tests;
* Demonstrating negative HIV, HBsAg and HCV-Ab screen tests;
* With mild-to-moderate persistent asthma for at least 6 months prior to Screening, and having used inhaled β-agonist(s) for asthma control;
* Demonstrating a Mean Screening Baseline FEV1 at 50.0 - 85.0 % of predicted normal;
* Demonstrating a ≥ 15.0% Airway Reversibility in FEV1 within 30(±5) min after inhaling 2 actuations of Proventil-HFA;
* Demonstrating Peak Inspiratory Flow Rate within 80-150 L/min;
* Demonstrating proficiency in the use of DPI and MDI after training;
* Females of child-bearing potential must be non-pregnant, non-lactating, and practicing a clinically acceptable form of birth control;
* Having properly consented to participate in the trial.

Exclusion Criteria:

* Smoking history of ≥ 10 pack-years, or having smoked within 6 months prior to Screening;
* Upper respiratory tract infections within 2 wk, or lower respiratory tract infection within 4 wk;
* Asthma exacerbations that required emergency care or hospitalized treatment, within 4 wk prior;
* Any current or recent respiratory conditions that might significantly affect pharmacodynamic response to the study drugs, besides asthma;
* Concurrent clinically significant cardiovascular, hematological, renal, neurologic, hepatic, endocrine, psychiatric, malignancies, or other illnesses that could impact on the conduct, safety and evaluation of the study;
* Known intolerance or hypersensitivity to any of the ingredients of the A006 or Proventil-HFA;
* Use of prohibited drugs or failure to observe the drug washout restrictions;
* Having been on other clinical drug/device studies in the last 30 days;
* Having donated blood within the last 30 days prior to Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Bronchodilatory efficacy after the escalating and cumulative-doses, up to 1,440 mcg. | -15 min predose, 15 min post dose 1, 2 and 3 and 15, 45, 90, 120, 180, 240, 360 min post dose 4
  Area Under the Curve (AUC)0-t of percent change in Forced Expiratory Volume in 1 second (FEV1), which is defined as the area under curve of post-dose FEV1 percentage changes from the Pre-dose Baseline FEV1 (FEV10) versus time. Doses are at 0, 30, 60 and 90 min.

SECONDARY OUTCOMES:
AUC0-t of change in FEV1 | -15, 15 min post 1, 2, and 3, and 15, 90, 120, 240, and 360min post dose 4
  AUC of FEV1 volume post-dose changes (change in Volume) from the Pre-dose Baseline FEV1 (FEV10). Doses are at 0, 30, 60 and 90 min.
Time to onset | 0 - 120 min
  Time to onset of bronchodilatory effect, determined by linear interpolation as the point where FEV1 % change first reaches ≥ 12% from FEV10.
Peak Response | 15 min post dose 1, 2 and 3 and 15, 45, 90, 120, 180, 240, and 360 min post dose 4
  The peak bronchodilator response, defined as the maximum post-dose FEV1 % change. Doses are at time 0, 30, 60, and 90 min.
Adverse Events | Time 0, 15, 45, 75, 105, 150, 195, 130, 190, 250, 435 minutes post dose 1
  The adverse drug events (ADE) that are observed with Proventil-HFA may be expected with the use of A006
Blood Analysis | -15, 10, 25,40, 55, 70, 85, 95, 115, 145, 175, 210, 270, 330, 690 min post dose 1
  serum glucose and potassium analysis and PK analysis
Vital Signs and Electrocardiogram (ECG) | -15, 5, 35, 65, 100, 155, 275, 455, 815 min post dose 1
  vital signs, including pulse and blood pressure and 12-lead ECG

CONTACTS AND LOCATIONS:
Overall Officials: Safety Monitor, Study Director — Amphastar Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - Amphastar Site 0025, Medford, Oregon
  - Amphastar Site 0026, Portland, Oregon
  - Amphastar Site 0032, San Antonio, Texas
  - Amphastar Site 0034, Seattle, Washington

REFERENCES:
- [Background] Ahrens RC. The role of the MDI and DPI in pediatric patients: "Children are not just miniature adults". Respir Care. 2005 Oct;50(10):1323-8; discussion 1328-30. PMID 16185368
- [Background] Goldstein DA, Tan YK, Soldin SJ. Pharmacokinetics and absolute bioavailability of salbutamol in healthy adult volunteers. Eur J Clin Pharmacol. 1987;32(6):631-4. doi: 10.1007/BF02456001. PMID 3653233
- [Background] Hindle M, Newton DA, Chrystyn H. Dry powder inhalers are bioequivalent to metered-dose inhalers. A study using a new urinary albuterol (salbutamol) assay technique. Chest. 1995 Mar;107(3):629-33. doi: 10.1378/chest.107.3.629. PMID 7874928
- [Background] Miller MR, Crapo R, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. General considerations for lung function testing. Eur Respir J. 2005 Jul;26(1):153-61. doi: 10.1183/09031936.05.00034505. No abstract available. PMID 15994402
- [Background] Pellegrino R, Viegi G, Brusasco V, Crapo RO, Burgos F, Casaburi R, Coates A, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson DC, MacIntyre N, McKay R, Miller MR, Navajas D, Pedersen OF, Wanger J. Interpretative strategies for lung function tests. Eur Respir J. 2005 Nov;26(5):948-68. doi: 10.1183/09031936.05.00035205. No abstract available. PMID 16264058
- [Background] Crapo RO, Morris AH, Gardner RM. Reference spirometric values using techniques and equipment that meet ATS recommendations. Am Rev Respir Dis. 1981 Jun;123(6):659-64. doi: 10.1164/arrd.1981.123.6.659. PMID 7271065
- [Background] Crapo RO, Morris AH, Clayton PD, Nixon CR. Lung volumes in healthy nonsmoking adults. Bull Eur Physiopathol Respir. 1982 May-Jun;18(3):419-25. PMID 7074238